CLINICAL TRIAL: NCT02548364
Title: Multicentric, Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Effect of Vitamin D on Ventricular Remodeling in Patients With Acute Myocardial Infarction
Brief Title: Effect of Vitamin D on Ventricular Remodeling in Patients With Acute Myocardial Infarction (VITDAMI)
Acronym: VITDAMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other); Spanish Society of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FJD-VITDAMI-14-01
Record Dates: First submitted 2015-07-06; First posted 2015-09-14 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Myocardial Infarction
Keywords: Vitamin D; Myocardial Infarction; Ventricular remodeling; Biomarkers
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling | interventions — Calcifediol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcifediol (Experimental): One capsule with 15,690 IU p.o. every two weeks
  Interventions: Drug: Calcifediol
- Placebo (Placebo Comparator): One capsule with placebo p.o. every two weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcifediol — calcifediol treatment
  Other Names: vitamin D
  Arms: Calcifediol
Drug: Placebo — placebo control group
  Arms: Placebo

SUMMARY:
To study the effect of calcifediol on left ventricular remodeling, mineral metabolism, plasma levels of several prognostic biomarkers and on endothelial function after an anterior myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years and maximum 85 years.
* Anterior myocardial infarction
* Sign informed consent

Exclusion Criteria:

* Death during the index event
* Age younger than 40 or older than 85 years
* Previous Infarction
* More than 7 days in hospitalization
* Systemic inflammatory or autoimmune disease
* Concomitant disorders limiting survival
* Concomitant cardiomyopathy
* Left ventricular hypertrophy > 16mm in females and > 17mm in males
* eGFR<45
* LVEF<30
* Incomplete revascularization
* Valvular prosthesis
* Aortic stenosis with mean gradient> 25 mmHg
* Moderate or severe valvular regurgitation
* Hypersensitivity or intolerance vitamin D supplement o excipient
* Blood Calcium >10.5 mg/dl
* Inability to follow.
* Difficulty in treatment compliance
* Contraindication for MRI, including indication to place a cardiac device
* Indication of therapy with vitamin D. Patient desires to take vitamin D.
* Drugs or conditions that interfere with the pharmacokinetics of calcifediol

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-10; Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Change in cardiac remodeling by MRI | 1 year
  It is a composite outcome measure. It will be analyzed by measuring the following parameters: myocardium at risk, size of infarcted myocardium, saved myocardium, ejection fraction, left ventricular telesystolic and telediastolic volumes

SECONDARY OUTCOMES:
Change in echocardiographic parameters | 1year
  It is a composite outcome measure. It will be analyzed by measuring the following parameters: ventricular thickness and diameters, contractility abnormalities, ejection fraction.
Change in mineral metabolism parameters | 1 year
  It is a composite outcome measure. It will be analyzed by measuring plasma levels of calcidiol, FGF-23, klotho, phosphate, and PTH
Change in prognostic biomarkers levels | 1 year
  It is a composite outcome measure. It will be analyzed by measuring plasma levels of NT-proBNP, hsCRP, MCP-1 and galectin-3
Change in lipid levels | 1 year
  It is a composite outcome measure. It will be analyzed by measuring plasma levels of TC, LDL, HDL, TG and non-HDL Cholesterol
Change in flow mediated vasodilation | 1 year
Adverse event rate | 1.5, 3, 6, 9, 12 and 13 months
% of treatment compliance | 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: JOSE TUÑON, MD, PhD, Principal Investigator — IIS-FJD
Locations (7):
- Spain (7):
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Hospital de Móstoles, Móstoles, Madrid
  - Hospital Infanta Elena, Valdemoro, Madrid
  - Fundación Jiménez Díaz, Madrid

REFERENCES:
- [Derived] Tunon J, Gonzalez-Hernandez I, Llanos-Jimenez L, Alonso-Martin J, Escudier-Villa JM, Tarin N, Cristobal C, Sanz P, Pello AM, Acena A, Carda R, Orejas M, Tomas M, Beltran P, Calero Rueda M, Marcos E, Serrano-Antolin JM, Gutierrez-Landaluce C, Jimenez R, Cabezudo J, Curcio A, Peces-Barba G, Gonzalez-Parra E, Munoz-Siscart R, Gonzalez-Casaus ML, Lorenzo A, Huelmos A, Goicolea J, Ibanez B, Hernandez G, Alonso-Pulpon LM, Farre J, Lorenzo O, Mahillo-Fernandez I, Egido J. Design and rationale of a multicentre, randomised, double-blind, placebo-controlled clinical trial to evaluate the effect of vitamin D on ventricular remodelling in patients with anterior myocardial infarction: the VITamin D in Acute Myocardial Infarction (VITDAMI) trial. BMJ Open. 2016 Aug 5;6(8):e011287. doi: 10.1136/bmjopen-2016-011287. PMID 27496232